CLINICAL TRIAL: NCT06930690
Title: Dexamethasone for Ureteral STent Symptoms (DUSTS): A Randomized, Double-blinded Controlled Study
Brief Title: Dexamethasone for Ureteral STent Symptoms (DUSTS)
Acronym: DUSTS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Monica Morgan, Assistant Professor of Clinical Urology, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00037902
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Ureteral Stent-Related Symptom
Keywords: Ureteral Stent; Nephrolithiasis; Ureteral Stent Discomfort; Ureteral Stent-Related Symptom
MeSH Terms: conditions — Nephrolithiasis | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Dexamethasone 20 mg
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection
- Control Arm (Active Comparator): Dexamethasone 4 mg
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate Injection — One time dose of dexamethasone sodium phosphate given intravenously at the time of surgery

SUMMARY:
The purpose of this study to learn if high-dose dexamethasone, a type of long-acting steroid, works to decrease urinary symptoms and pain after ureteroscopy and stent placement for kidney stones. The main question it aims to answer is:

1) Does high-dose steroid change the quality of life score on day 2 after surgery

Researchers will compare high-dose of dexamethasone (20 mg) to a standard dose of dexamethasone (4 mg) to see if a higher dose of the drug will help with urinary symptoms and pain

Participants will:

1. randomly receive 20 mg or 4 mg of dexamethasone (20 mg) at the time of surgery
2. fill out a questionnaire day 1 and day 2 after surgery
3. fill out a medication diary for one week after surgery
4. visit the clinic on day 2 after surgery for checkup
5. visit the clinic on day 4-7 after surgery for check up

DETAILED DESCRIPTION:
Patient will be in the study for a duration of 30 days. Randomization will be performed on the day of surgery using the NIH Clinical Trial Randomization Tool.

In the preoperative area, a finger stick blood glucose (FSBG) level will be checked. Patients with a FSBG ≥126 mg/dL will be disqualified from the study.

Following induction of general anesthesia, the anesthesiologist will administer the study drug (dexamethasone 20 mg vs 4 mg) without members of the surgery team in the operating room. This is the only treatment that will be done for research purpose. The following are part of routine clinical care. Perioperative antibiotic prophylaxis will be given by the discretion of the surgeon following Houston Methodist Hospital (HMH) and American Urological Association (AUA) guidelines. Ureteroscopy (URS) will then be performed. If laser lithotripsy will be performed, a holmium or thulium laser will be used. After URS is completed, a ureteral stent will be placed. The length of the stent will be determined by the patient's height. Stent string can be left on or removed prior to placement based on surgeon discretion. Subjects will be prescribed tamsulosin (0.4 mg, #30), docusate (100 mg, #60), extended-release oxybutynin (10 mg, #30), and tramadol (50 mg, #20) OR acetaminophen/codeine (325/30 mg, #20). Stent removal will be performed in clinic 4-7 days after surgery.

FSBG will be checked upon patient's arrival to the PACU. Postop corrective insulin lispro LOW dose will be administered if needed and FSBG will be rechecked in one hour according to Houston Methodist's "Diabetes and Hyperglycemia Management Postop" protocol.

Persistent hyperglycemia will be defined as FSBG ≥200 one hour after insulin administration. If patient is experiencing persistent hyperglycemia, they will be admitted for monitoring. An endocrinologist will be consulted for evaluation and treatment of hyperglycemia and its acute complication if suspected.

Patients will be observed in the PACU for at least 3 hours. After meeting standard discharge criteria, a final FSBG will be checked. Patients will only be discharged if FSBG is between 81 mg/dL and 200 mg/dL.

For research purposes, the Ureteral Stent Symptom Questionnaire (USSQ) is a validated questionnaire that will be used to assess and measure ureteral stent symptoms in this study. One set of the USSQ will be given to patients as a packet after surgery, and patients will be instructed to take the questionnaire on POD 1. Subjects will be telephoned by study staff on POD1 to maximize the completion rate of forms and will be inquired if they have signs and symptoms of DKA/HHS (e.g. polyuria, polydipsia, fruity breath odor, nausea, vomiting, abdominal pain). Subjects will be instructed to seek care at the nearest emergency room if needed, preferably Houston Methodist Hospital.

Subjects will also be given a medication diary to record the use of all medication prescribed following surgery. Opioid use will be converted to total morphine equivalents.

Patients will also be instructed to follow up on POD2 in the clinic for a nursing visit and with the study coordinator. The second set of USSQ will be given and patients will fill out the questionnaire in the office. During this visit, a random FSBG will also be checked for research purpose. If FSBG ≥200 mg/dL, patients will be directed to seek care at the emergency room at Houston Methodist Hospital. An endocrinologist will be consulted for evaluation and treatment of hyperglycemia and its acute complication if suspected.

Patient will come to the clinic again on POD4-7 for stent removal. Subjects will not fill out the USSQ questionnaire on these days. The medication diary will be collected from the subjects during this visit. A random FSBG will also be performed during this follow up visit for research purpose. If FSBG ≥200 mg/dL, patients will be directed to seek care at the emergency room at Houston Methodist Hospital. An endocrinologist will be consulted for evaluation and treatment of hyperglycemia and its acute complication if suspected.

On the 30 day after their surgery, subjects will be telephone by study staff to record any adverse events including side effects, emergency room visits, or hospital admission. Their electronic medical records within the 30 days will also be reviewed by the study team.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old
2. Patients who are undergoing unilateral retrograde ureteroscopy (semi-rigid or flexible) with planned ureteral stent placement for treatment of renal/ureteral stones
3. Patients who can read and understand English
4. Patients who can follow up post-operatively within 7 days at Houston Methodist Hospital

Exclusion Criteria:

1. Untreated UTI
2. HbA1c ≥6.5 on preoperative testing
3. Patients with prior diagnosis of any type of diabetes mellitus
4. Patients with immunosuppression, including chronic corticosteroid use
5. Patients with bleeding disorder
6. Patients with chronic liver disease, cirrhosis, and liver failure.
7. Patients taking strong CYP3A4 inducers or inhibitors within two weeks of screening
8. Chronic opioid analgesic use
9. Congenital renal abnormalities (e.g. pelvic kidney, ureteric duplication) that may impair stent placement
10. Concurrent genitourinary malignancy
11. Urinary diversion
12. Renal transplantation
13. History of interstitial cystitis/painful bladder syndrome, prostatitis, pelvic pain due to other conditions (e.g. endometriosis)
14. Neurologic disorder (e.g. spinal cord injury, multiple sclerosis, spina bifida)
15. Pregnant or breastfeeding
16. Patients with cognitive impairments or untreated psychiatric illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Global Quality of Life Score of Ureteral Stent Symptom Questionnaire (USSQ) | Day 2 after surgery
  A 1 to 7 rating scale used to measure survey participants' feeling if they were advised to have another stent inserted, from 1 = delighted to 7 = terrible.

SECONDARY OUTCOMES:
Urinary Index Score of the USSQ | Day 2 after surgery
  This domain assesses urinary symptoms (e.g., urgency, frequency, dysuria) and consists of multiple questions, each answered using a Likert-type scale.
  Higher scores indicate greater symptom severity.
Pain Index Score of the USSQ | Day 2 after surgery
  This domain assesses pain (e.g., flank pain, suprapubic discomfort) and consists of multiple questions, each answered using a Likert-type scale.
  Higher scores indicate greater symptom severity.
General Health Index Score of the USSQ | Day 2 after surgery
  This domain assesses general health (overall health perception and well-being) and consists of multiple questions, each answered using a Likert-type scale.
  Higher scores indicate greater symptom severity.
Work Performance Index Score of the USSQ | Day 2 after surgery
  This domain assesses work performance (impact of stent symptoms on work productivity) and consists of multiple questions, each answered using a Likert-type scale.
  Higher scores indicate greater symptom severity.
Opioid Use After Surgery | From intervention to stent removal at 4-7 days after surgery
  The amount of of prescribed opioid (in morphine equivalent dose) used during the time subjects have their stent in situ

OTHER OUTCOMES:
Incidence of steroid-related adverse events | Within 30 days
  Incidence of the steroid-induced hyperglycemia (SIHG) as defined as random blood glucose ≥200 mg/dL and hyperglycemia-related adverse events including diabetic ketoacidosis (DKA) and hyperosmolar syndrome (HHS)
Incidence of UTIs | Within 30 days
  Incidence of symptomatic urinary tract infections (UTIs)
Number of ER visit or hospital admission | Within 30 days
  Number of unplanned emergency room visit or hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Monica Morgan, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No